CLINICAL TRIAL: NCT05859503
Title: A Comparison Study of the Perclose Proglide (TM) SMC System Versus Figure-of-8- Suture Technique for Closure of Large-bore Femoral Venous Access. (PERCLOSE-PROGLIDE)
Brief Title: A Comparison Study of the Perclose Proglide (TM) SMC System Versus Figure-of-8- Suture Technique for Closure of Large-bore Femoral Venous Access.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PERCLOSE PROGLIDE
Record Dates: First submitted 2023-05-03; First posted 2023-05-16 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Diseases
Keywords: Femoral venous access closure techniques; Figure-of-8 suture,Perclose-Proglide system
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perclose-Proglide system
  Interventions: Other: Closure Strategy with Perclose-Proglide system
- Figure-of-8
  Interventions: Other: Closure Strategy with figure-of-8

INTERVENTIONS:
Other: Closure Strategy with Perclose-Proglide system — Patients who have required Perclose-Proglide system in Percutaneous Interventional Procedure
  Groups: Perclose-Proglide system
Other: Closure Strategy with figure-of-8 — Patients who have required the manual compression with figure-of-8 in Percutaneous Interventional Procedure
  Groups: Figure-of-8

SUMMARY:
This study aims to compare the efficacy and safety of two strategies for closing large caliber venous access in patients undergoing percutaneous procedures: compression with figure-of-8 suture versus closure with the Perclose-Proglide system.

DETAILED DESCRIPTION:
This is a retrospective observational study that aims to compare two strategies for closing large-caliber femoral venous access in patients who have undergone percutaneous procedures.

The study's goal is to determine if there are significant differences in terms of efficacy and safety between the two closure strategies. Figure-of-8 suture compression is a well-established technique that has been used for decades to close large-bore femoral venous access, while the Perclose-Proglide system is a relatively new medical device that could have great utility for the closure of large-bore femoral venous access. By comparing these two strategies, researchers hope to determine the safety and effectiveness of the Perclose-Proglide system for closing large-bore femoral venous access in patients undergoing percutaneous procedures.

ELIGIBILITY:
Inclusion Criteria:

Patients will meet all inclusion criteria:

* Adult patients aged > 18 years
* Patients who have undergone percutaneous interventional procedures
* Patients in whom the procedures have been performed with femoral venous access
* Patients who have required large caliber pods ≥ 14 French.

Exclusion Criteria:

Patients must not meet any exclusion criteria:

* Patients who have required access with surgical exposure.
* Patients who have required ipsilateral arterial access with a large caliber ≥ 14 French
* Patients with previous vascular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone interventional procedures and who have required the use of figure-of-8 suture versus Perclose-Proglide system closure
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Major vascular complications | 30 days
  Incidence of patients with Major vascular complications
Assessment of Major vascular complications | Discharge (assessed up to day 5)
  Incidence of patients with Major vascular complications
Assessment of rebleeding | Discharge (assessed up to day 5)
  Incidence of patients with rebleeding
Rebleeding | 30 days
  Incidence of patients with rebleeding

SECONDARY OUTCOMES:
Assessment of Death | Discharge (assessed up to day 5)
  Incidence of dead patients
Assessment of Death | 30 days
  Incidence of dead patients
Assessment of Death related to vascular access | 30 days
  Incidence of dead patients related to vascular access
Assessment of Death related to vascular access | Discharge (assessed up to day 5)
  Incidence of dead patients related to vascular access
Assessment of Hematoma | 24 hours
  Incidence of patients with hematoma the venous puncture
Assessment of Hematoma Size | 24 hours
  Area in cm of the hematoma at the venous puncture in patients with hematoma
Assessment of Vascular access point infection | Discharge (assessed up to day 5)
  Incidence of patients with infection in vascular access point
Assessment of Vascular access point infection | 30 days
  Incidence of patients with infection in vascular access point
Assessment of Urinary infections | 30 days
  Incidence of patients with urinary infection
Assessment of Urinary infections | Discharge (assessed up to day 5)
  Incidence of patients with urinary infection
Assessment of sitting-walking time | Discharge (assessed up to day 5)
  Time in hours between the patient sitting and walking after the vascular access
Assessment of Technical success | 1 minute after closure performed
  Technical success when complete hemostasis is less than 1 minute after closure strategy performed
Assessment of Clinical success | Discharge (assessed up to day 5)
  Technical success in the absence of events after closure strategy

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall D'Hebron, Barcelona, Spain

REFERENCES:
- [Background] Hamid T, Rajagopal R, Pius C, Clarke B, Mahadevan VS. Preclosure of large-sized venous access sites in adults undergoing transcatheter structural interventions. Catheter Cardiovasc Interv. 2013 Mar;81(4):586-90. doi: 10.1002/ccd.24358. Epub 2012 Nov 8. PMID 22431302
- [Background] Jensen CJ, Schnur M, Lask S, Attanasio P, Gotzmann M, Kara K, Hanefeld C, Mugge A, Wutzler A. Feasibility of the Figure-of-8-Suture as Venous Closure in Interventional Electrophysiology: One Strategy for All? Int J Med Sci. 2020 Apr 6;17(7):965-969. doi: 10.7150/ijms.42593. eCollection 2020. PMID 32308550
- [Background] Mohanty S, Trivedi C, Beheiry S, Al-Ahmad A, Horton R, Della Rocca DG, Gianni C, Gasperetti A, Abdul-Moheeth M, Turakhia M, Natale A. Venous access-site closure with vascular closure device vs. manual compression in patients undergoing catheter ablation or left atrial appendage occlusion under uninterrupted anticoagulation: a multicentre experience on efficacy and complications. Europace. 2019 Jul 1;21(7):1048-1054. doi: 10.1093/europace/euz004. PMID 30726903
- [Background] Pracon R, Bangalore S, Henzel J, Cendrowska-Demkow I, Pregowska-Chwala B, Tarnowska A, Dzielinska Z, Chmielak Z, Witkowski A, Demkow M. A randomized comparison of modified subcutaneous "Z"-stitch versus manual compression to achieve hemostasis after large caliber femoral venous sheath removal. Catheter Cardiovasc Interv. 2018 Jan 1;91(1):105-112. doi: 10.1002/ccd.27003. Epub 2017 Mar 17. PMID 28303670
- [Background] Geis NA, Pleger ST, Chorianopoulos E, Muller OJ, Katus HA, Bekeredjian R. Feasibility and clinical benefit of a suture-mediated closure device for femoral vein access after percutaneous edge-to-edge mitral valve repair. EuroIntervention. 2015 Mar;10(11):1346-53. doi: 10.4244/EIJV10I11A231. PMID 24694560
- [Background] Noori VJ, Eldrup-Jorgensen J. A systematic review of vascular closure devices for femoral artery puncture sites. J Vasc Surg. 2018 Sep;68(3):887-899. doi: 10.1016/j.jvs.2018.05.019. Epub 2018 Jun 29. PMID 30146036